CLINICAL TRIAL: NCT04832191
Title: 1.3 Role of Contrast-enhanced Mammography and Dynamic Contrast-enhanced MRI in the Assessment of Solid Breast Lesions
Brief Title: CE-MRI&CESM in Solid Breast Lesions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Basma Fawzy Mohamed Gad El-Rab, Assistant professor, Assiut University
Other Study IDs: CE-MRI&CESM in breast lesions
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Breast Neoplasms
Keywords: CE-SM /CE-MRI/solid breast lesions
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: CE-SM — contrast enhanced spectral mammography &contrast enhanced magnetic resonance imaging
  Other Names: CE-MRI

SUMMARY:
Our study aimed to assess the accuracy of CE-SM in comparison to contrast-enhanced breast MRI in the evaluation of solid breast lesions.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women, responsible for 23% of cancer in females worldwide (1).

Early detection and accurate diagnosis of breast cancer aims to reduce morbidity and mortality and have essential role in management and improved prognosis of breast cancer (2).

Mammography has been established as the imaging modality for screening and early detection of breast cancer; however, it is accused of having low sensitivity and specificity in women with dense breasts (3).

Contrast-enhanced MRI considered the gold standard method for diagnosis of breast cancer; but, it has many limitations as high cost, long examination time and limited availability (4,5).

Contrast-enhanced spectral mammogram (CESM) is considered now a relatively new imaging modality which can provide both anatomic and functional information of the breast lesion similar to MRI (6).

CESM like contrast-enhanced MRI (CE-MRI) is used to detect angiogenesis of the lesion in the mammography suite. It includes high- and low-energy images during a single compression after contrast injection (7).

The advantage of CESM over MRI is that it is less expensive and easier to perform with shorter examination time. Also, the higher sensitivity of MRI is plagued by numerous false-positive foci of enhancement (8).

Also, CESM can replace MRI in case of patient contraindicating for MRI as patients with pacemakers, aneurysm clips or metal implants, or severe claustrophobia (7).

So, our study aims to determine the value of CESM and answer the question of does CESM could replace CE-MRI in diagnosing breast cancer? so,our study aimed to assess the accuracy of CESM in comparison to contrast-enhanced breast MRI in the evaluation of solid breast lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have previously undergone mammography (MG) and ultrasound and have a solid (BIRADs III and more) breast lesion.

Exclusion Criteria:

* Cystic breast lesions
* BIRADs I and II breast lesions(benign)
* Pregnancy
* History of allergic reaction to iodinated contrast agent
* Renal insufficiency
* Other contraindications to MRI include pacemaker, claustrophobia or metal prosthesis.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presented clinically with solid breast lesions.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
comparison between accuracy of CESM and CE-MRI in diagnosing breast cancer. | baseline
  Measurement of sensitivity, specificity and predictive values of CESM and CE-MRI in diagnosing breast cancer.

REFERENCES:
- [Background] Zhu X, Huang JM, Zhang K, Xia LJ, Feng L, Yang P, Zhang MY, Xiao W, Lin HX, Yu YH. Diagnostic Value of Contrast-Enhanced Spectral Mammography for Screening Breast Cancer: Systematic Review and Meta-analysis. Clin Breast Cancer. 2018 Oct;18(5):e985-e995. doi: 10.1016/j.clbc.2018.06.003. Epub 2018 Jun 15. PMID 29983379
- [Background] Li L, Roth R, Germaine P, Ren S, Lee M, Hunter K, Tinney E, Liao L. Contrast-enhanced spectral mammography (CESM) versus breast magnetic resonance imaging (MRI): A retrospective comparison in 66 breast lesions. Diagn Interv Imaging. 2017 Feb;98(2):113-123. doi: 10.1016/j.diii.2016.08.013. Epub 2016 Sep 26. PMID 27687829